CLINICAL TRIAL: NCT03067389
Title: Evaluation of a Combined Breast Cancer Risk Derived From a Polygenic Risk Score and the Tyrer-Cuzick Model
Brief Title: Combined Breast Cancer Risk Study
Status: Completed | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HCP-018
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Hereditary Cancer
MeSH Terms: interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- History of invasive breast cancer: Subjects with a diagnosis of invasive breast cancer within the past 12 months will provide a blood or saliva sample for genetic diagnostic testing and provide information about their personal medical and cancer history and family cancer history.
  Interventions: Diagnostic Test: Diagnostic test
- No history of invasive breast cancer: Subjects with no history of breast cancer will provide a blood or saliva sample for genetic diagnostic testing and provide information about their personal medical and cancer history and family cancer history.
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Genetic diagnostic test

SUMMARY:
A prospective, non-interventional study in women 18 to 84 years of age. Subjects will provide a sample for genetic testing and information about their medical and family history. The results of the genetic test will be combined with clinical data to validate a method of predicting breast cancer risk.

DETAILED DESCRIPTION:
This is a prospective, non- interventional study. Women presenting at imaging centers for routine breast cancer screening or breast cancer diagnostic assessment and who provide written informed consent will undergo genetic testing. Subjects will also provide information about their personal medical and cancer history and family cancer history. The results of the genetic test will be combined with the subject's clinical information, family history, and a risk assessment model to validate a new method of predicting breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Women without breast cancer:

* 18 to 84 years of age
* Western/Northern European, Central/Eastern European, or Ashkenazi ancestry
* No history of invasive breast cancer

Women with a history of breast cancer:

* 18 to 84 years of age
* Western/Northern European, Central/Eastern European, or Ashkenazi ancestry
* Pathologically confirmed invasive breast cancer diagnosed within the past 12 months

Exclusion Criteria:

* Unwilling to provide written informed consent
* Women with history of ductal carcinoma in situ (DCIS).
* Patient has had a prior breast biopsy, exclusive of a breast biopsy diagnostic of breast cancer, that showed either hyperplasia, atypical hyperplasia, lobular carcinoma in situ (LCIS), or the specific histologic result is unknown to the patient

Ages: 18 Years to 84 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women presenting at imaging centers for a breast cancer diagnostic assessment visit or preventative screening visit.
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2016-02-06 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate that a combined breast cancer risk derived from a polygenic risk score and a breast cancer risk assessment model is a better predictor of breast cancer than the risk assessment model alone | Baseline

SECONDARY OUTCOMES:
To derive a distribution of polygenic risk scores in an unselected patient population | baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Holmsn, MD, Study Director — Myriad Genetics, Inc.
Locations (4):
- United States (4):
  - The Breast Center of Northwest Arkansas, Fayetteville, Arkansas
  - Bethesda Health, Boynton Beach, Florida
  - Cuda Women's Health Center, Hyannis, Massachusetts
  - Elizabeth Wende Breast Care, Rochester, New York

IPD SHARING:
Plan to Share IPD: No